CLINICAL TRIAL: NCT02255383
Title: Persona The Personalized Knee System TKA Outcomes Study: Prospective Multicenter Study of the Persona Knee System
Brief Title: Persona Total Knee Arthroplasty Outcomes Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSU2014-02K
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2024-11

CONDITIONS: Knee Pain Chronic; Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Polyarthritis; Moderate Varus, Valgus or Flexion Deformities; Avascular Necrosis of the Femoral Condyle
Keywords: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Polyarthritis; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis; Genu Valgum | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PERSONA TKA (Other): Primary total knee arthroplasty subjects that receive the Zimmer Persona Total Knee System
  Interventions: Device: Zimmer Persona Total Knee System

INTERVENTIONS:
Device: Zimmer Persona Total Knee System — Primary Total Knee Arthroplasty
  Other Names: Total Knee Arthroplasty; Total Knee Replacement

SUMMARY:
The primary objective of this study is to obtain implant survivorship and clinical outcomes data for commercially available Persona fixed bearing knee implants used in total knee arthroplasty. The assessment will include implant survivorship and clinical performance.

DETAILED DESCRIPTION:
The study design is a prospective, multicenter, study of the commercially available Persona fixed bearing knee implants. The study will require each site to obtain IRB approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

All study subjects will undergo preoperative clinical evaluations prior to their total knee arthroplasty. The post-operative clinical and radiographic evaluations will be conducted at 6 weeks, 6 months, 1 year, 2, 3, 5, 7, and 10 years.

The primary objective of this study is to obtain implant survivorship and clinical outcomes data for the commercially available Persona fixed bearing implants used in primary total knee arthroplasty. The assessments will include: implant survivorship based on removal of a study device; safety based on incidence and frequency of adverse events; and clinical performance measured by overall pain and function, quality of life data, radiographic parameters and survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18-75 years of age, inclusive
* Patient qualifies for primary total knee arthroplasty based on physical exam and medical history, including diagnosis of severe knee pain and disability due to at least one of the following: a) rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis; b) collagen disorders and/or avascular necrosis of the femoral condyle; c) post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy; d) moderate valgus, varus, or flexion deformities; or e) the salvage of previously failed surgical attempts that did not include partial or total knee arthroplasty of the ipsilateral knee
* Patient has participated in a study-related Informed Consent process
* Patient is willing and able to provide written Informed Consent by signing and dating the IRB or EC approved Informed Consent Form
* Patient is willing and able to complete scheduled study procedures and follow-up evaluations
* Independent of study participation, patient is a candidate for commercially available Persona fixed bearing knee components implanted in accordance with product labeling

Exclusion Criteria:

* Patient is currently participating in any other surgical intervention studies or pain management studies
* Previous history of infection in the affected joint and/or other local/systemic infection that may affect the prosthetic joint
* Insufficient bone stock on femoral or tibial surfaces
* Skeletal immaturity
* Neuropathic arthropathy
* Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb
* Stable, painless arthrodesis in a satisfactory functional position
* Severe instability secondary to the absence of collateral ligament integrity
* Rheumatoid arthritis accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin
* Patient has a known or suspected sensitivity or allergy to one or more of the implant materials
* Patient is pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.)
* Patient has previously received partial or total knee arthroplasty for the ipsilateral knee

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2014-07; Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | 10 years
  Knee Society Score

SECONDARY OUTCOMES:
EQ-5D | 10 years
  EQ-5D

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Colorado Joint Replacement, Denver, Colorado
  - Orthopaedic & Spine Center of the Rockies, Fort Collins, Colorado
  - Denver-Vail Orthopedics, Parker, Colorado
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Henry County Orthopedics and Sports Medicine, New Castle, Indiana
  - UNC Department of Orthopaedics, Chapel Hill, North Carolina
  - OrthoCarolina, Charlotte, North Carolina
  - Raleigh Orthopaedic Clinic, Raleigh, North Carolina
  - Lindner Research Center, Cincinnati, Ohio
  - SportsMedicine Grant & Orthopaedic Associates, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Tennessee Orthopaedic Foundation for Education and Research, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Jordan Young Institute, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No